CLINICAL TRIAL: NCT05286021
Title: Comparison of the Clinical Performance and Safety of the Ambu®AuraGainTM Laryngeal Mask in Children Undergoing Surgery in the Supine and Prone Position - A Prospective, Noninferiority Clinical Trial
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2021-0079
Record Dates: First submitted 2022-03-06; First posted 2022-03-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2022-03

CONDITIONS: Bone Marrow Examination; Urologic Surgical Procedures; Orthopedic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supine group: Children undergoing surgery in the supine position using the Ambu Auragain
- Prone group: Children undergoing surgery in the prone position using the Ambu Auragain

SUMMARY:
The Ambu Auragain is a 2nd generation laryngeal mask airway that is widely used in adult and pedicatric patients. While its use is generally recommended in patients undergoing surgery in the supine position, depending on patient characteristics, type of surgery and experience of the anesthesiologist, it may also be used in the lateral or prone position. There have been reports of LMA use in patients undergoing short procedures in the prone position, but its safety in pediatric patients is not clear. This study was designed to compare oropharyngeal leak pressure between children undergoing surgery in the supine and prone position using the Ambu Auragain LMA.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients undergoing surgery within 2 hours under general anesthesia in either the supine or prone position using the Ambu Auragain LMA.

Patients aged 2-12 years, weight 10-30 kg, ASA class 1~3

Exclusion Criteria:

Active URI, symptomatic lung disease (uncontrolled asthma, pneumonia etc), patients with history of difficult airway, anticipated difficult mask ventilation, risk of aspiration such as gastroesophageal reflux

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will be done in pediatric patients between the ages 2 and 12 years, weight 10 and 30 kg, that are eligible to use the Ambu Auragain LMA for surgical procedures within 2 hours. The patients will undergo surgery in either the supine or prone position.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure immediately after LMA insertion | During procedure (Immediately after AmbuAuragain LMA insertion)
  Oropharyngeal leak pressure is commonly used as a parameter to assess the clinical performance of supraglottic airway devices (SADs). It is defined as the anesthesia circuit pressure at which a gas leak occurs around the SAD.

SECONDARY OUTCOMES:
Oropharyngeal leak pressure 10 minutes after positioning for surgery | 10 minutes after positioning (either supine or prone position) for surgery.
  Oropharyngeal leak pressure is commonly used as a parameter to assess the clinical performance of supraglottic airway devices (SADs). It is defined as the anesthesia circuit pressure at which a gas leak occurs around the SAD.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No